CLINICAL TRIAL: NCT03141112
Title: The Benefits of Early Initiation of Continuous Renal Replacement Therapy (CRRT) in Patients With Severe Sepsis
Brief Title: The Benefits of Early Initiation of Continual Renal Replacement Therapy in Patients With Severe Sepsis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Radovan Uvizl (Other)
Responsible Party: Sponsor-Investigator, Radovan Uvizl, MUDr., University Hospital Olomouc
Organization: University Hospital Olomouc (Other)
Other Study IDs: ECRRT 51/16
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis | interventions — Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- early CRRT initiation: Patients in ICU with severe sepsis, both gender, adult, over 18 years od age. Initiation of renal replacement therapy up to 48 hours after reaching criteria of severe sepsis.
  Interventions: Procedure: renal replacement therapy
- late CRRT initiation: Patients in ICU with severe sepsis, both gender, adult, over 18 years od age. Initiation of renal replacement therapy after 48 hours after reaching criteria of severe sepsis.
  Interventions: Procedure: renal replacement therapy

INTERVENTIONS:
Procedure: renal replacement therapy

SUMMARY:
The study will evaluate the benefit of early initiation of CRRT in the initial phase of severe sepsis in patients admitted to the ICU. Primary evaluated end-point is 28-day mortality. Secondarily evaluated end-point is length of ICU-stay, length of stay in hospital, duration of mechanical ventilation. There are two groups. One group of participants with early CRRT initiation and another group with late CRRT initiation. Reference group no CRRT.

DETAILED DESCRIPTION:
The aim is to determine the optimal timing of initiation of CRRT with respect to the degree and duration of acute kidney injury (AKI) in ICU patients. The CRRT parameters and the duration of therapy will be monitored, depending on initial biochemical and clinical values of the patient. Part of the study is the follow-up of patients with a 3-month delay.

ELIGIBILITY:
Inclusion Criteria:

* reaching criteria of severe sepsis, ICU admission

Exclusion Criteria:

* pregnant women, younger than 18 years, reaching contraindications for initiation of renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in severe sepsis (reaching criteria for severe sepsis), both gender, age over 18 years old, admisset in ICU.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 days
  yes/no

SECONDARY OUTCOMES:
duration of mechanical ventilation | 28 days
  days of mechanical ventilation including weening

OTHER OUTCOMES:
length of stay | 3 months
  length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Radovan Uvizl, Principal Investigator — UH Olomouc, Czech Republic

IPD SHARING:
Plan to Share IPD: Undecided